CLINICAL TRIAL: NCT01386281
Title: Drug Use Investigation of Julina Tablets 0.5 mg (Postmenopausal Osteoporosis)
Brief Title: Julina Post-marketing Surveillance for Climacteric Symptoms in Japan
Acronym: JULINA-CLIMA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15073
Record Dates: First submitted 2011-06-16; First posted 2011-07-01 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Julina; Postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: E2 transdermal (Julina, BAY86-5435)

INTERVENTIONS:
Drug: E2 transdermal (Julina, BAY86-5435) — Patients in daily life treatment receiving Julina for postmenopausal osteoporosis

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Julina for postmenopausal osteoporosis. The objective of this study is to assess safety and efficacy of using Julina in clinical practice. A total 100 patients will be recruited and followed 3 years since starting Julina administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Julina for postmenopausal osteoporosis

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who have received a prescription of Julina on the basis of the decision of the treating gynecologist. The study is expected to collect data of 100 patients in about 20 gynecological practices in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subject who received Julina | After Julina administration, upto 1 year

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation with baseline data (such as demographic data, concomitant disease) and dose of Julina | At baseline and after Julina administration, upto 1 year
Change from baseline in grad of hot flush and sweating at the end of Julina treatment | At baseline and at end of Julina treatment, upto 1 year
Change from baseline in with/without vaginal atrophy at the end of Julina treatment | At baseline and at end of Julina treatment, upto 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan